CLINICAL TRIAL: NCT02575508
Title: A Phase Ib/II Study of BGJ398 in Combination Modified FOLFIRINOX in Treatment-Naïve Metastatic Pancreatic Cancer Patients
Brief Title: Pan FGFR Kinase Inhibitor BGJ398 and Combination Chemotherapy in Treating Patients With Untreated Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: drug supply issues
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 265214; NCI-2015-01597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 265214 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Colon Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Rectal Adenocarcinoma; Stage III Pancreatic Cancer; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IV Pancreatic Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms | interventions — Fluorouracil; dehydroftorafur; Irinotecan; Oxaliplatin; infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (oxaliplatin, irinotecan, fluorouracil, BGJ398) (Experimental): Patients receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously over 46 hours on days 1 and 15. Patients also receive pan FGFR kinase inhibitor BGJ398 PO QD on days 8-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Drug: pan FGFR Kinase Inhibitor BGJ398; Other: Pharmacological Study

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: pan FGFR Kinase Inhibitor BGJ398 — Given IV
  Other Names: BGJ398
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of pan fibroblast growth factor receptor (FGFR) kinase inhibitor BGJ398 when given together with fluorouracil, irinotecan hydrochloride and oxaliplatin (combination chemotherapy) in treating patients with untreated pancreatic cancer that has spread to another place in the body. Pan FGFR kinase inhibitor BGJ398 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil, irinotecan hydrochloride and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pan FGFR kinase inhibitor BGJ398 together with fluorouracil, irinotecan hydrochloride and oxaliplatin may be a better treatment for pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine dose-limiting toxicity, the maximum tolerated dose and recommended phase II dose of BGJ398 (pan FGFR kinase inhibitor BGJ398) administered in combination with modified (m)FOLFIRINOX (fluorouracil, irinotecan hydrochloride and oxaliplatin) in patients with advanced pancreatic and colorectal cancer patients. (Phase Ib)

II. To determine the 6-month overall survival rate of patients with treatment-naïve metastatic pancreatic ductal adenocarcinoma treated with BGJ398 plus mFOLFIRINOX. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic profile of BGJ398, fluorouracil, oxaliplatin, irinotecan (irinotecan hydrochloride) and their metabolites when administered in combination and explore for drug-drug interactions. (Phase Ib)

II. To determine the 1-year overall survival rate, response rate, progression free survival and cancer antigen (CA)19-9 changes in treatment-naïve metastatic pancreatic cancer patients treated with BGJ398 plus mFOLFIRINOX. (Phase II)

III. To determine the safety and tolerability of BGJ398 in combination with mFOLFIRINOX in the study population.

IV. To explore plasma and tumor biomarkers associated with efficacy to the study combination.

OUTLINE: This is a phase Ib, dose-escalation study of pan FGFR kinase inhibitor BGJ398 followed by a phase II study.

Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously over 46 hours on days 1 and 15. Patients also receive pan FGFR kinase inhibitor BGJ398 orally (PO) once daily (QD) on days 8-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days and then every 4 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase Ib: Histologically or cytologically confirmed adenocarcinoma of the pancreas, colon or rectum which disease is advanced (defined as not surgically curable) or metastatic in whom combination treatment using fluorouracil, oxaliplatin and irinotecan is a rational option
* All patients must consent to provide archival tumor samples; non-availability of evaluable tumor samples does not exclude patient from the study
* Phase II: Patients with histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma that have not received systemic chemotherapy for advanced or metastatic disease; the definitive diagnosis of metastatic pancreatic adenocarcinoma will be made by integrating the histopathological data within the context of the clinical and radiographic data
* Phase II: The initial 20 patients must have evaluable baseline tumor samples; evaluable samples are defined as those obtained by core biopsy or surgical resection and amendable to histological analysis; samples obtained by fine needle aspiration biopsy are not considered evaluable; patients who do not have evaluable archival tumor samples must consent to a tumor core biopsy prior to starting study treatment and, patients who consent to the baseline tumor biopsy will be eligible to receive study treatment irrespective of whether the samples obtained are evaluable
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Phase Ib: Have evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Phase II: Have at least 1 metastatic lesion other than the primary pancreatic tumor that is evaluable per RECIST 1.1 criteria; lesions previously irradiated are not considered evaluable
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (International System of Units [SI] units 1.5 x 10^9/L)
* Platelets >= 100,000 cells/mm^3 (SI units 100 x 10^9/L)
* Hemoglobin >= 9.0 g/dL (SI units 90 g/L)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x ULN; in patients with known hepatic involvement, AST and ALT =< 5 x ULN are allowed
* Serum creatinine =< 1.5 x ULN or estimated creatinine clearance >= 60 mL/min by the Cockcroft-Gault equation
* International normalized ratio (INR) =< 1.5
* Inorganic phosphorus =< ULN
* Ionized calcium =< ULN
* Ability to swallow and retain oral medication
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Phase II: Patient who recurs with metastatic disease =< 6 months of completing adjuvant chemotherapy after curative-intent surgical resection is not eligible; patients who recur with metastatic disease > 6 months after completion of adjuvant chemotherapy are eligible
* Phase II: Patients that previously received systemic chemotherapy for metastatic or advanced pancreatic adenocarcinoma are not eligible
* Phase II: Diagnosis of any second malignancy within the last 3 years except for adequately treated basal cell carcinoma, or squamous cell skin carcinoma or in-situ cervical carcinoma
* Patients with clinically significant ascites requiring paracentesis on 2 or more occasions within 4 weeks prior to start of study treatment
* Known hypersensitivity to BGJ398, fluorouracil, oxaliplatin, irinotecan or to any of the excipients
* Homozygous UDP glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1)*28 (i.e. 7 TA repeats) gene alleles; the UGT1A1 test should be conducted per local institutional practice
* Palliative radiation treatment (e.g., pain control, bony lesions at risk of fracture) completed =< 2 weeks of starting study treatment; patient will be eligible if palliative radiotherapy is completed > 2 weeks from the start of study treatment and has recovered from radiotherapy toxicities
* Pulmonary embolus or thrombosis of the deep venous system (deep vein thrombosis [DVT]) within 2 weeks of starting study treatment; patients who had a history of thromboembolic disease should be stable on therapeutic anticoagulation using low molecular weight (LMW) heparin for at least 2 weeks prior to the start of study treatment; use of warfarin (or derivatives) is not allowed at the start of study treatment
* Patients with known symptomatic brain metastases requiring steroids and/or antiepileptic therapy; patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study treatment, and have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable; patients with leptomeningeal involvement are excluded
* Current evidence of corneal or retinal disorder/keratopathy including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, confirmed by ophthalmologic examination
* Prior FGFR inhibitor therapy
* History or current evidence of:

  * Tissue calcification including, but not limited to, the soft tissue, kidneys, intestines, myocardium and lung with the exception of calcified lymph nodes and asymptomatic coronary calcification
  * Endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc
* Patients who are currently receiving or consuming

  * Medications that are known strong inducers or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) =< 14 days of starting study treatment

    • Medications with a known risk of prolonging the QT interval or inducing Torsades de Pointes =< 7 days prior to start of study treatment
  * Amiodarone =< 180 days prior to start of study treatment
  * Grapefruit, grapefruit juice, pomegranates, star fruits, Seville oranges or products =< 7 days prior to start of study treatment
  * Warfarin (or derivatives)
* Uncontrolled intercurrent illness including, but not limited to,

  * Ongoing or active infection
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Clinically significant cardiac disease including any of the following:

    * Congestive heart failure requiring treatment (New York Heart Association grade >= 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi gated acquisition scan (MUGA) scan or echocardiogram
    * Uncontrolled hypertension (defined as systolic blood pressure [BP] >= 160 mmHg OR diastolic BP >= 100 mmHg despite maximal anti-hypertensive medications: refer to World Health Organization [WHO]-International Society of Hypertension [ISH] guidelines)
    * History or presence of clinically significant ventricular arrhythmias, atrial fibrillation, resting bradycardia, or conduction abnormality
    * Unstable angina pectoris or acute myocardial infarction < 3 months prior to starting study treatment
    * Corrected QT using the Fredericia's formula (QTcF) > 450 msec (males); > 470 msec (females)
    * History of congenital long QT syndrome
* Known (historical) positive human immunodeficiency virus (HIV) serology, active hepatitis B, or active hepatitis C infection
* Major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury =< 4 weeks and minor procedures (including percutaneous biopsies, placement of vascular access device, laparoscopy +/- biopsy) =< 1 week prior to starting study treatment; patients who have minor procedure(s) > 1 week prior to starting study treatment and have recovered from side effects of such procedure are eligible
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Pregnant or nursing women; a negative pregnancy test (serum or urine) =< 3 days prior to starting study treatment
* Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) unless they are using highly effective methods of contraception during study treatment and for 3 months following the discontinuation of study treatment; highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject); periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening); for female patients on the study the vasectomized male partner should be the sole partner for that patient
  * Combination of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository; oral contraceptives (OC), injected or implanted hormonal methods are not allowed as the sole method of contraception
* Post-menopausal women are allowed to participate in this study; women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse during and for 3 months after the last dose of the study treatment and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase Ib) | Up to 28 days
Maximum tolerated dose (MTD) and recommended phase II dose of BGJ398 in combination with mFOLFIRINOX, defined as the dose with a probability of DLT of 0.30 graded according to the NCI CTCAE version 4.0 (Phase Ib) | 28 days
  The MTD will be estimated using isotonic regression (cumulative cohort design).
Overall survival (Phase II) | Time from the start of the study treatment until death, last follow-up or drop-out, assessed at 6 months
  The overall survival will be summarized using Kaplan-Meier methods, from which an estimate of the 6-month survival rate and corresponding standard error will be obtained using the methods proposed by Breslow and Day.

SECONDARY OUTCOMES:
Changes in CA19-9 expression levels (Phase II) | Baseline to 2 years
  The CA19-9 expression will be reported by time as mean, median, standard deviation, and percentiles. Changes in expression will be evaluated using the paired t-test or Wilcoxon signed rank test, as appropriate.
Incidence of adverse events graded according to the NCI CTCAE version 4.0 | Up to 28 days after completion of study treatment
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles. The frequency of toxicities will also be tabulated for the dose estimated to be the MTD and RP2D in phase Ib.
Objective tumor response (Phase II) | Up to 2 years
  The objective tumor responses will be reported as frequencies and relative frequencies, with the response rates estimated with Clopper-Pearson 95% confidence intervals.
Progression free survival (Phase II) | Up to 2 years
  The progression free survival will be summarized using standard Kaplan-Meier methods, with estimates of median survival and given survival rates (i.e., 1 year) will be obtained with 95% confidence intervals.
Potential associations between response rate and tumor biomarkers (Phase II) | Up to 2 years
  Will be evaluated using logistic regression models and associated exact methods.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States